CLINICAL TRIAL: NCT03689049
Title: SPIDER: A Structured Process Informed by Data, Evidence and Research - A Research and Quality Improvement Collaboration Supporting Practices in Improving Care for Complex Elderly Patients
Brief Title: SPIDER: A Research & QI Collaboration Supporting Practices in Improving Care for Complex Elderly Patients
Acronym: SPIDER
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto Practice Based Research Network (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Toronto (Other); North York General Hospital (Other); College of Family Physicians of Canada (Other); University of Ottawa (Other); University of Alberta (Other); University of Calgary (Other); University of Manitoba (Other); Research Manitoba (Other); Fonds de la Recherche en Santé du Québec (Other Government); Université de Montréal (Other); Nova Scotia Health Authority (Other); Dalhousie University (Other); Dalhousie Medical Research Foundation (Unknown); Doctors Nova Scotia (Unknown); Memorial University of Newfoundland (Other); University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KPG-156886
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Polypharmacy; Inappropriate Prescribing; Aged; Primary Health Care; Quality Improvement; Electronic Health Records
Keywords: Polypharmacy; Deprescribing; Aged Adult; Elderly Patient; Primary Health Care; Quality Improvement; Practice Facilitation; Learning Collaborative; Electronic Medical Records (EMR)

STUDY DESIGN:
Intervention Model Description: The intervention will first be tested for feasibility using a single-arm, prospective, explanatory mixed approach. What we learn from the feasibility will then be applied to a 2-arm pragmatic cluster RCT where practices enrolled in the intervention group will be compared with those enrolled in the usual care group. Randomization will be at the practice level to avoid potential contamination where physicians practicing at the same location are enrolled in different arms.
Masking Description: Blinding of participants cannot be achieved in pragmatic trials of QI interventions in primary care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPIDER (Experimental): QI Learning Collaboratives.
  Interventions: Procedure: SPIDER; Procedure: Usual Care
- Usual Care (Placebo Comparator): Standard primary care.
  Interventions: Procedure: Usual Care

INTERVENTIONS:
Procedure: SPIDER — The SPIDER intervention will include a family physician-led inter-professional practice team participating in 3-4 Learning Collaboratives over a period of 12 months, reviewing validated and comparable practice EMR data and working with a QI Coach to develop strategies and implement changes to improve care for elderly patients living with complex care needs and taking ten or more unique medications.
  Arms: SPIDER
Procedure: Usual Care — Physicians and their teams enrolled in this arm will follow the best scientific evidence available to provide standard care that is in the best interest of their patients.

SUMMARY:
Elders living with multiple chronic conditions often take many drugs (polypharmacy); some of the drugs may not benefit them or may be harmful. The Canadian Institute for Health Information has reported that about one-quarter of Canadian seniors are prescribed ten or more different drugs each year. Polypharmacy can result in poorer health, reduced quality of life and high healthcare costs. Choosing Wisely Canada and the Canadian Deprescribing Network have suggested wiser uses for the following four Potentially Inappropriate Prescriptions (PIPs): drugs that reduce stomach acid; reduce anxiety and induce sleep; treat agitation; and treat type 2 diabetes but have a high risk of low blood sugar. To improve care for elderly patients living with polypharmacy, we propose SPIDER: a Structured Process Informed by Data, Evidence and Research. Using quality improvement (QI) and supported by Electronic Medical Record (EMR) data, SPIDER will invite family doctors, nurses, pharmacists and front desk staff to participate in Learning Collaboratives and learn from each other. The practice teams will work with a QI Coach to identify areas to improve, develop strategies and implement changes tailored to the local practice context. The objective of this study is to determine whether SPIDER will reduce PIPs for patients 65 years or older who are on ten or more different drugs. The study will also explore patient experience and provider satisfaction with SPIDER and assess the cost of running SPIDER. The study will first be tested for feasibility in Toronto, Edmonton and Montreal. Findings will then guide a Randomized Controlled Trial (RCT) in Calgary, Winnipeg, Ottawa, Montreal and Halifax where practices enrolled in the SPIDER intervention will be compared with those in usual care.

DETAILED DESCRIPTION:
Polypharmacy is pervasive amongst elderly patients living with multiple chronic conditions and the prevalence is increasing. The Canadian Institute for Health Information recently reported that 26.5% Canadian seniors were prescribed ten or more different drugs in 2016. A member of our team (S. Dahrouge) has found that number of prescription proved to be the most reliable index of persistent complexity and high cost in patients 65 years or older. There is also an association between number of prescription and potentially inappropriate prescriptions (PIPs). Analyses conducted on 86 practices affiliated with the University of Toronto Practice Based Research Network (UTOPIAN) have found that family physicians look after a mean of 24 older patients prescribed ten or more medications each year. Polypharmacy in the elderly is associated with elevated risks of adverse drug reactions, frailty and falls. It also increases healthcare, drug, and hospitalization costs. While several medications can be problematic, the following four classes of PIPs have been specifically identified by Choosing Wisely Canada and the Canadian Deprescribing Network as targets for wiser uses in elders: proton pump inhibitors (PPIs), sedative hypnotics such as benzodiazepines, antipsychotics for agitation and medications with a higher risk of hypoglycemia such as long-acting sulfonylureas. To improve care for elderly patients living with polypharmacy, we propose SPIDER: a Structured Process Informed by Data, Evidence and Research. Leveraging existing Quality Improvement (QI) capacity and provision of validated EMR data, SPIDER will engage inter-professional practice teams. They will participate in Learning Collaboratives and work with QI Coaches to identify areas of improvement, develop strategies and implement changes to improve care. The study aims to assess whether SPIDER can reduce PIPs in older patients prescribed ten or more medications. Patient experience, provider satisfaction and cost-effectiveness of SPIDER will also be evaluated. The study will first be tested for feasibility in Toronto, Edmonton and Montreal. Findings will then guide a pragmatic cluster RCT in Calgary, Winnipeg, Ottawa, Montreal and Halifax where practices enrolled in the SPIDER intervention will be compared with those in usual care.

ELIGIBILITY:
Inclusion criteria:

1. At practice level: a) contributes EMR data to the repository of a Practice Based Research Network (PBRN) that participates in CPCSSN; and b) includes a primary care provider (PCP) who consents to participate and lead the practice QI team.
2. At PCP level: a) practices comprehensive family medicine in an office setting (academic or non-academic); and b) consents to participate and allow the research staff to provide study information to their eligible patients.
3. At patient level: a) 65 years or older; b) has at least one office visit during the past 2 years; and c) has received ten or more different prescription medications (as indicated in the EMR) in the past year.

Exclusion criteria:

1. At practice level: a) Does not use EMR; b) does not contributes EMR data to the repository of a PBRN that participates in CPCSSN; or c) none of the PCPs at the practice consents to participate.
2. At PCP level: a) does not practice comprehensive family medicine in an office setting; b) does not consent to participate; c) does not allow the research staff to contact or provide study information to their eligible patients; or d) has left the practice.
3. At patient level: a) younger than 65 years of age; b) has not visited a practice over the past 2 years; or c) has received fewer than ten different prescription medications in the past year.

(Note:

* PBRN: Practice Based Research Network;
* CPCSSN: the Canadian Primary Care Sentinel Surveillance Network)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2018-03-26 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of Potentially Inappropriate Prescriptions (PIPs). | 12 months
  The primary outcome is the number of prescribed medications identified as one of the four targeted PIPs recommended by Choosing Wisely Canada and the Canadian DePrescribing Network (CaDeN).

SECONDARY OUTCOMES:
Patient perception of SPIDER | 12 months
  Qualitative methods (survey and interview) will be used to measure patients' perception of SPIDER. Patients' attitude toward polypharmacy and deprescribing will be measured using a survey adopted from Veterans Affairs Multi-dimensional Survey. Patients' experience with the process, symptoms, relationship with the care provider, empowerment and care coordination dimension will be measured using an interview.
Care provider perception of SPIDER | 12 months
  Qualitative methods (survey and focus group) will be used to measure care providers' perception of SPIDER, including the dimensions of acceptability, implementation, adaptation, integration, practicality and efficacy.
Cost-utility of SPIDER | 12 months
  The cost-utility of SPIDER will be measured as the incremental gain in quality of life (measured by EuroQol-5D) between the two arms in relation to intervention costs and by comparing the differences in investments and healthcare costs captured through EMR data and emergency room use and hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Greiver, MD, Principal Investigator — North York General Hospital
Locations (9):
- Canada (9):
  - Southern Alberta Primary Care Research Network (SAPCReN), Calgary, Alberta
  - Northern Alberta Primary Care Research Network (NAPCReN), Edmonton, Alberta
  - British Columbia node of the pan-Canadian CPCSSN (BC-CPCSSN), Vancouver, British Columbia
  - Manitoba Primary Care Research Network (MaPCReN), Winnipeg, Manitoba
  - Atlantic Practice Based Research Network (APBRN), St. John's, Newfoundland and Labrador
  - Maritime Family Practice Research Network (MaRNet-FP), Halifax, Nova Scotia
  - Ottawa Practice Enhancement Network (OPEN ), Ottawa, Ontario
  - University of Toronto Practice Based Research Network, Toronto, Ontario
  - Réseau de recherche en soins primaires de l'Université de Montréal (RRSPUM), Laval, Quebec

IPD SHARING:
Plan to Share IPD: Yes
This study uses some data from the Canadian Primary Care Sentinel Surveillance Network (CPCSSN) for outcome measurement. A data dictionary is available from CPCSSN. While data sharing agreements prohibit CPCSSN from making the data publicly available, access may be granted to those who meet pre-specified criteria for confidential access, available at http://cpcssn.ca/research-resources/cpcssn-data-for-research/; researchers with additional questions can contact CPCSSN by using the link. Outcome data collected for this project can be made available to researchers upon request; a SPIDER study member will need to be part of the new work to ensure adequate interpretation of the data. The study protocol including statistical analysis plan and informed consent form will be publicly available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 12 months of study completion
Access Criteria: Outcome data collected for this project can be made available to researchers upon request; a SPIDER study member will need to be part of the new work to ensure adequate interpretation of the data.

REFERENCES:
- [Background] Berk ML, Monheit AC, Hagan MM. How the U.S. spent its health care dollar: 1929-1980. Health Aff (Millwood). 1988 Fall;7(4):46-60. doi: 10.1377/hlthaff.7.4.46. No abstract available. PMID 3147235
- [Background] Berk ML, Monheit AC. The concentration of health expenditures: an update. Health Aff (Millwood). 1992 Winter;11(4):145-9. doi: 10.1377/hlthaff.11.4.145. PMID 1483633
- [Background] Riley GF. Long-term trends in the concentration of Medicare spending. Health Aff (Millwood). 2007 May-Jun;26(3):808-16. doi: 10.1377/hlthaff.26.3.808. PMID 17485760
- [Background] Blumenthal D, Causino N, Chang YC, Culpepper L, Marder W, Saglam D, Stafford R, Starfield B. The duration of ambulatory visits to physicians. J Fam Pract. 1999 Apr;48(4):264-71. PMID 10229250
- [Background] Rais S, Nazerian A, Ardal S, Chechulin Y, Bains N, Malikov K. High-cost users of Ontario's healthcare services. Healthc Policy. 2013 Aug;9(1):44-51. PMID 23968673
- [Background] Chang HY, Boyd CM, Leff B, Lemke KW, Bodycombe DP, Weiner JP. Identifying Consistent High-cost Users in a Health Plan: Comparison of Alternative Prediction Models. Med Care. 2016 Sep;54(9):852-9. doi: 10.1097/MLR.0000000000000566. PMID 27326548
- [Background] Hochman M, Asch SM. Disruptive Models in Primary Care: Caring for High-Needs, High-Cost Populations. J Gen Intern Med. 2017 Apr;32(4):392-397. doi: 10.1007/s11606-016-3945-2. Epub 2017 Feb 27. PMID 28243870
- [Background] Berk ML, Monheit AC. The concentration of health care expenditures, revisited. Health Aff (Millwood). 2001 Mar-Apr;20(2):9-18. doi: 10.1377/hlthaff.20.2.9. PMID 11260963
- [Background] Guilcher SJ, Bronskill SE, Guan J, Wodchis WP. Who Are the High-Cost Users? A Method for Person-Centred Attribution of Health Care Spending. PLoS One. 2016 Mar 3;11(3):e0149179. doi: 10.1371/journal.pone.0149179. eCollection 2016. PMID 26937955
- [Background] Tanuseputro P, Wodchis WP, Fowler R, Walker P, Bai YQ, Bronskill SE, Manuel D. The health care cost of dying: a population-based retrospective cohort study of the last year of life in Ontario, Canada. PLoS One. 2015 Mar 26;10(3):e0121759. doi: 10.1371/journal.pone.0121759. eCollection 2015. PMID 25811195
- [Background] Lavan AH, Gallagher P. Predicting risk of adverse drug reactions in older adults. Ther Adv Drug Saf. 2016 Feb;7(1):11-22. doi: 10.1177/2042098615615472. PMID 26834959
- [Background] Reeve E, Ong M, Wu A, Jansen J, Petrovic M, Gnjidic D. A systematic review of interventions to deprescribe benzodiazepines and other hypnotics among older people. Eur J Clin Pharmacol. 2017 Aug;73(8):927-935. doi: 10.1007/s00228-017-2257-8. Epub 2017 Apr 30. PMID 28456823
- [Background] Fletcher PC, Berg K, Dalby DM, Hirdes JP. Risk factors for falling among community-based seniors. J Patient Saf. 2009 Jun;5(2):61-6. doi: 10.1097/PTS.0b013e3181a551ed. PMID 19920442
- [Background] Tannenbaum C, Martin P, Tamblyn R, Benedetti A, Ahmed S. Reduction of inappropriate benzodiazepine prescriptions among older adults through direct patient education: the EMPOWER cluster randomized trial. JAMA Intern Med. 2014 Jun;174(6):890-8. doi: 10.1001/jamainternmed.2014.949. PMID 24733354
- [Background] Lindblad CI, Hanlon JT, Gross CR, Sloane RJ, Pieper CF, Hajjar ER, Ruby CM, Schmader KE, Multidisciplinary Consensus Panel. Clinically important drug-disease interactions and their prevalence in older adults. Clin Ther. 2006 Aug;28(8):1133-1143. doi: 10.1016/j.clinthera.2006.08.006. PMID 16982290
- [Background] Gurwitz JH, Field TS, Harrold LR, Rothschild J, Debellis K, Seger AC, Cadoret C, Fish LS, Garber L, Kelleher M, Bates DW. Incidence and preventability of adverse drug events among older persons in the ambulatory setting. JAMA. 2003 Mar 5;289(9):1107-16. doi: 10.1001/jama.289.9.1107. PMID 12622580
- [Background] Barry HE, Cooper JA, Ryan C, Passmore AP, Robinson AL, Molloy GJ, Darcy CM, Buchanan H, Hughes CM. Potentially Inappropriate Prescribing Among People with Dementia in Primary Care: A Retrospective Cross-Sectional Study Using the Enhanced Prescribing Database. J Alzheimers Dis. 2016 Apr 11;52(4):1503-13. doi: 10.3233/JAD-151177. PMID 27079714
- [Background] Hovstadius B, Petersson G. The impact of increasing polypharmacy on prescribed drug expenditure-a register-based study in Sweden 2005-2009. Health Policy. 2013 Feb;109(2):166-74. doi: 10.1016/j.healthpol.2012.09.005. Epub 2012 Nov 26. PMID 23195435
- [Background] Akazawa M, Imai H, Igarashi A, Tsutani K. Potentially inappropriate medication use in elderly Japanese patients. Am J Geriatr Pharmacother. 2010 Apr;8(2):146-60. doi: 10.1016/j.amjopharm.2010.03.005. PMID 20439064
- [Background] Morgan SG, Hunt J, Rioux J, Proulx J, Weymann D, Tannenbaum C. Frequency and cost of potentially inappropriate prescribing for older adults: a cross-sectional study. CMAJ Open. 2016 Jun 22;4(2):E346-51. doi: 10.9778/cmajo.20150131. eCollection 2016 Apr-Jun. PMID 27398383
- [Background] Steinberg M, Lyketsos CG. Atypical antipsychotic use in patients with dementia: managing safety concerns. Am J Psychiatry. 2012 Sep;169(9):900-6. doi: 10.1176/appi.ajp.2012.12030342. PMID 22952071
- [Background] Pollock K, Grime J. The cost and cost-effectiveness of PPIs--GP perspectives and responses to a prescribing dilemma and their implications for the development of patient-centred healthcare. Eur J Gen Pract. 2003 Dec;9(4):126-33, 140. doi: 10.3109/13814780309160421. PMID 14733400
- [Background] Wang PS, Schneeweiss S, Avorn J, Fischer MA, Mogun H, Solomon DH, Brookhart MA. Risk of death in elderly users of conventional vs. atypical antipsychotic medications. N Engl J Med. 2005 Dec 1;353(22):2335-41. doi: 10.1056/NEJMoa052827. PMID 16319382
- [Background] Farrell B, Pottie K, Thompson W, Boghossian T, Pizzola L, Rashid FJ, Rojas-Fernandez C, Walsh K, Welch V, Moayyedi P. Deprescribing proton pump inhibitors: Evidence-based clinical practice guideline. Can Fam Physician. 2017 May;63(5):354-364. PMID 28500192
- [Background] Hogan DB, Maxwell CJ, Fung TS, Ebly EM; Canadian Study of Health and Aging. Prevalence and potential consequences of benzodiazepine use in senior citizens: results from the Canadian Study of Health and Aging. Can J Clin Pharmacol. 2003 Summer;10(2):72-7. PMID 12879145
- [Background] Wang PS, Bohn RL, Glynn RJ, Mogun H, Avorn J. Zolpidem use and hip fractures in older people. J Am Geriatr Soc. 2001 Dec;49(12):1685-90. doi: 10.1111/j.1532-5415.2001.49280.x. PMID 11844004
- [Background] Tannenbaum C, Farrell B, Shaw J, Morgan S, Trimble J, Currie J, Turner J, Rochon P, Silvius J. An Ecological Approach to Reducing Potentially Inappropriate Medication Use: Canadian Deprescribing Network. Can J Aging. 2017 Mar;36(1):97-107. doi: 10.1017/S0714980816000702. Epub 2017 Jan 16. PMID 28091333
- [Background] Garfinkel D, Ilhan B, Bahat G. Routine deprescribing of chronic medications to combat polypharmacy. Ther Adv Drug Saf. 2015 Dec;6(6):212-33. doi: 10.1177/2042098615613984. PMID 26668713
- [Background] Thompson W, Hogel M, Li Y, Thavorn K, O'Donnell D, McCarthy L, Dolovich L, Black C, Farrell B. Effect of a Proton Pump Inhibitor Deprescribing Guideline on Drug Usage and Costs in Long-Term Care. J Am Med Dir Assoc. 2016 Jul 1;17(7):673.e1-4. doi: 10.1016/j.jamda.2016.04.020. Epub 2016 Jun 8. PMID 27289201
- [Background] Page AT, Clifford RM, Potter K, Schwartz D, Etherton-Beer CD. The feasibility and effect of deprescribing in older adults on mortality and health: a systematic review and meta-analysis. Br J Clin Pharmacol. 2016 Sep;82(3):583-623. doi: 10.1111/bcp.12975. Epub 2016 Jun 13. PMID 27077231
- [Background] Iyer S, Naganathan V, McLachlan AJ, Le Couteur DG. Medication withdrawal trials in people aged 65 years and older: a systematic review. Drugs Aging. 2008;25(12):1021-31. doi: 10.2165/0002512-200825120-00004. PMID 19021301
- [Background] Jansen J, Naganathan V, Carter SM, McLachlan AJ, Nickel B, Irwig L, Bonner C, Doust J, Colvin J, Heaney A, Turner R, McCaffery K. Too much medicine in older people? Deprescribing through shared decision making. BMJ. 2016 Jun 3;353:i2893. doi: 10.1136/bmj.i2893. No abstract available. PMID 27260319
- [Background] Boulin M, Diaby V, Tannenbaum C. Preventing Unnecessary Costs of Drug-Induced Hypoglycemia in Older Adults with Type 2 Diabetes in the United States and Canada. PLoS One. 2016 Sep 20;11(9):e0162951. doi: 10.1371/journal.pone.0162951. eCollection 2016. PMID 27648831
- [Background] Farrell B, Black C, Thompson W, McCarthy L, Rojas-Fernandez C, Lochnan H, Shamji S, Upshur R, Bouchard M, Welch V. Deprescribing antihyperglycemic agents in older persons: Evidence-based clinical practice guideline. Can Fam Physician. 2017 Nov;63(11):832-843. PMID 29138153
- [Background] Schmader KE, Hanlon JT, Pieper CF, Sloane R, Ruby CM, Twersky J, Francis SD, Branch LG, Lindblad CI, Artz M, Weinberger M, Feussner JR, Cohen HJ. Effects of geriatric evaluation and management on adverse drug reactions and suboptimal prescribing in the frail elderly. Am J Med. 2004 Mar 15;116(6):394-401. doi: 10.1016/j.amjmed.2003.10.031. PMID 15006588
- [Background] Spinewine A, Swine C, Dhillon S, Lambert P, Nachega JB, Wilmotte L, Tulkens PM. Effect of a collaborative approach on the quality of prescribing for geriatric inpatients: a randomized, controlled trial. J Am Geriatr Soc. 2007 May;55(5):658-65. doi: 10.1111/j.1532-5415.2007.01132.x. PMID 17493184
- [Background] Herxheimer A, McGettigan P. Problems of polypharmacy. BMJ. 2013 Dec 23;347:f7500. doi: 10.1136/bmj.f7500. No abstract available. PMID 24366533
- [Background] Frank C, Weir E. Deprescribing for older patients. CMAJ. 2014 Dec 9;186(18):1369-76. doi: 10.1503/cmaj.131873. Epub 2014 Sep 2. No abstract available. PMID 25183716
- [Background] Lenander C, Elfsson B, Danielsson B, Midlov P, Hasselstrom J. Effects of a pharmacist-led structured medication review in primary care on drug-related problems and hospital admission rates: a randomized controlled trial. Scand J Prim Health Care. 2014 Dec;32(4):180-6. doi: 10.3109/02813432.2014.972062. Epub 2014 Oct 27. PMID 25347723
- [Background] Bokhof B, Junius-Walker U. Reducing Polypharmacy from the Perspectives of General Practitioners and Older Patients: A Synthesis of Qualitative Studies. Drugs Aging. 2016 Apr;33(4):249-66. doi: 10.1007/s40266-016-0354-5. PMID 26915076
- [Background] Birtwhistle R, Keshavjee K, Lambert-Lanning A, Godwin M, Greiver M, Manca D, Lagace C. Building a pan-Canadian primary care sentinel surveillance network: initial development and moving forward. J Am Board Fam Med. 2009 Jul-Aug;22(4):412-22. doi: 10.3122/jabfm.2009.04.090081. PMID 19587256
- [Background] Mold JW, Peterson KA. Primary care practice-based research networks: working at the interface between research and quality improvement. Ann Fam Med. 2005 May-Jun;3 Suppl 1(Suppl 1):S12-20. doi: 10.1370/afm.303. PMID 15928213
- [Background] Thorpe KE, Zwarenstein M, Oxman AD, Treweek S, Furberg CD, Altman DG, Tunis S, Bergel E, Harvey I, Magid DJ, Chalkidou K. A pragmatic-explanatory continuum indicator summary (PRECIS): a tool to help trial designers. CMAJ. 2009 May 12;180(10):E47-57. doi: 10.1503/cmaj.090523. Epub 2009 Apr 16. No abstract available. PMID 19372436
- [Background] Schwartz D, Lellouch J. Explanatory and pragmatic attitudes in therapeutical trials. J Chronic Dis. 1967 Aug;20(8):637-48. doi: 10.1016/0021-9681(67)90041-0. No abstract available. PMID 4860352
- [Background] Boutron I, Moher D, Altman DG, Schulz KF, Ravaud P; CONSORT Group. Extending the CONSORT statement to randomized trials of nonpharmacologic treatment: explanation and elaboration. Ann Intern Med. 2008 Feb 19;148(4):295-309. doi: 10.7326/0003-4819-148-4-200802190-00008. PMID 18283207
- [Background] Campbell MK, Piaggio G, Elbourne DR, Altman DG; CONSORT Group. Consort 2010 statement: extension to cluster randomised trials. BMJ. 2012 Sep 4;345:e5661. doi: 10.1136/bmj.e5661. No abstract available. PMID 22951546
- [Background] Brehaut JC, Colquhoun HL, Eva KW, Carroll K, Sales A, Michie S, Ivers N, Grimshaw JM. Practice Feedback Interventions: 15 Suggestions for Optimizing Effectiveness. Ann Intern Med. 2016 Mar 15;164(6):435-41. doi: 10.7326/M15-2248. Epub 2016 Feb 23. PMID 26903136
- [Background] Linsky A, Simon SR, Stolzmann K, Meterko M. Patient Perceptions of Deprescribing: Survey Development and Psychometric Assessment. Med Care. 2017 Mar;55(3):306-313. doi: 10.1097/MLR.0000000000000642. PMID 27579916
- [Background] Reeve E, To J, Hendrix I, Shakib S, Roberts MS, Wiese MD. Patient barriers to and enablers of deprescribing: a systematic review. Drugs Aging. 2013 Oct;30(10):793-807. doi: 10.1007/s40266-013-0106-8. PMID 23912674
- [Background] Turner JP, Edwards S, Stanners M, Shakib S, Bell JS. What factors are important for deprescribing in Australian long-term care facilities? Perspectives of residents and health professionals. BMJ Open. 2016 Mar 10;6(3):e009781. doi: 10.1136/bmjopen-2015-009781. PMID 26966056
- [Background] Sekhon M, Cartwright M, Francis JJ. Acceptability of healthcare interventions: an overview of reviews and development of a theoretical framework. BMC Health Serv Res. 2017 Jan 26;17(1):88. doi: 10.1186/s12913-017-2031-8. PMID 28126032
- [Background] Montiel-Luque A, Nunez-Montenegro AJ, Martin-Aurioles E, Canca-Sanchez JC, Toro-Toro MC, Gonzalez-Correa JA; Polipresact Research Group. Medication-related factors associated with health-related quality of life in patients older than 65 years with polypharmacy. PLoS One. 2017 Feb 6;12(2):e0171320. doi: 10.1371/journal.pone.0171320. eCollection 2017. PMID 28166266
- [Background] MacCarthy D, Kallstrom L, Kadlec H, Hollander M. Improving primary care in British Columbia, Canada: evaluation of a peer-to-peer continuing education program for family physicians. BMC Med Educ. 2012 Nov 9;12:110. doi: 10.1186/1472-6920-12-110. PMID 23140230
- [Background] Farrell B, Richardson L, Raman-Wilms L, de Launay D, Alsabbagh MW, Conklin J. Self-efficacy for deprescribing: A survey for health care professionals using evidence-based deprescribing guidelines. Res Social Adm Pharm. 2018 Jan;14(1):18-25. doi: 10.1016/j.sapharm.2017.01.003. Epub 2017 Jan 28. PMID 28214150
- [Background] Green LA, White LL, Barry HC, Nease DE Jr, Hudson BL. Infrastructure requirements for practice-based research networks. Ann Fam Med. 2005 May-Jun;3 Suppl 1(Suppl 1):S5-11. doi: 10.1370/afm.299. PMID 15928219
- [Background] Bello AK, Ronksley PE, Tangri N, Singer A, Grill A, Nitsch D, Queenan JA, Lindeman C, Soos B, Freiheit E, Tuot D, Mangin D, Drummond N. A national surveillance project on chronic kidney disease management in Canadian primary care: a study protocol. BMJ Open. 2017 Aug 4;7(8):e016267. doi: 10.1136/bmjopen-2017-016267. PMID 28780553
- [Background] Southgate D, Greiver M, Hubka G, Kostka K, Moineddin R, Moienedin M, Pencharz J, Bogetta H, Mazariegos C, Guindon JA, Petroff A. Effect of a Group Behavioural Management Program on Emotional Regulation of Food Choices: A Pilot Randomized Controlled Trial. Can J Diet Pract Res. 2017 Sep 1;78(3):137-140. doi: 10.3148/cjdpr-2017-006. Epub 2017 Mar 23. PMID 28333551
- [Background] Vickers AJ, Altman DG. Statistics notes: Analysing controlled trials with baseline and follow up measurements. BMJ. 2001 Nov 10;323(7321):1123-4. doi: 10.1136/bmj.323.7321.1123. No abstract available. PMID 11701584
- [Background] Udow-Phillips M, Ehrlich E, Kofke-Egger H. Health Care Cost Drivers: Chronic Disease, Comorbidity, and Health Risk Factors in the U.S. and Michigan | Center for Healthcare Research & Transformation. Ann Arbor: Center for Healthcare Research & Transformation 2010.
- [Background] Moturu S, Johnson W, Liu H. Predictive risk modelling for forecasting high-cost patients: A real-world application using Medicaid data. International Journal Biomedical Engineering and Technology. 2010;3(1-2):114-132.
- [Background] Wodchis W, Austin P, Newman A, Carollo A, Henry D. The Concentration of Health Care Spending: Little Ado (yet) About Much (money). 2012; https://www.cahspr.ca/en/presentation/5244423937dee8014beea024.
- [Background] Glazier R, Agha M, Creatore M, Gozdyra P. High Cost Health Care Users: A Focus on Health Links. 2017. http://www.torontohealthprofiles.ca/a_documents/aboutTheData/HealthQualityTablepresentationOnHighUsers.pdf.
- [Background] The Breakthrough Series: IHI's Collaborative Model for Achieving Breakthrough Improvement. IHI Innovation Series white paper. 2003. http://www.ihi.org/resources/Pages/IHIWhitePapers/TheBreakthroughSeriesIHIsCollaborativeModelforAchievingBreakthroughImprovement.aspx.
- [Background] Dahrouge S, Wodchis W. Identifying high users in Ontario - an algorithm for use in primary care practices. 2017;In press.
- [Background] Canadian Deprescribing Network: Deprescribing algorithms. 2017; https://www.deprescribingnetwork.ca/algorithms/.
- [Background] Donner A. Some aspects of the design and analysis of cluster randomization trials. Appl Stat. 1998;47:95-113.
- [Background] Romanow R. Building on values: the future of health care in Canada. Ottawa2002.
- [Background] Clement S. The self-efficacy expectations and occupational preferences of females and males. Journal of Occupational Psychology. 1987;60(3):257-265.
- [Background] Rosella LC, Fitzpatrick T, Wodchis WP, Calzavara A, Manson H, Goel V. High-cost health care users in Ontario, Canada: demographic, socio-economic, and health status characteristics. BMC Health Serv Res. 2014 Oct 31;14:532. doi: 10.1186/s12913-014-0532-2. PMID 25359294
- [Background] Wodchis W, Bushmeneva K, Nikitović M, McKillop IH, McKillop E. Guidelines on Person-level Costing Using Administrative Databases in Ontario. Working Paper Series. Vol 1. 2013.
- [Background] Wodchis WP, Austin PC, Henry DA. A 3-year study of high-cost users of health care. CMAJ. 2016 Feb 16;188(3):182-188. doi: 10.1503/cmaj.150064. Epub 2016 Jan 11. PMID 26755672
- [Background] WHO Collaborating Centre for drug statistic methodology - ATC/DDD Index. 2017; https://www.whocc.no/atc_ddd_index/.
- [Background] Greiver M, Martin K, Aliarzadeh B, Lambert-Lanning A, Leggett J. Implementing a scalable tool for quality improvement in primary care: a report for Canada Health Infoway. Toronto December 2013.
- [Background] Godwin M, Ruhland L, Casson I, MacDonald S, Delva D, Birtwhistle R, Lam M, Seguin R. Pragmatic controlled clinical trials in primary care: the struggle between external and internal validity. BMC Med Res Methodol. 2003 Dec 22;3:28. doi: 10.1186/1471-2288-3-28. PMID 14690550
- [Background] Garies S, Birtwhistle R, Drummond N, Queenan J, Williamson T. Data Resource Profile: National electronic medical record data from the Canadian Primary Care Sentinel Surveillance Network (CPCSSN). Int J Epidemiol. 2017 Aug 1;46(4):1091-1092f. doi: 10.1093/ije/dyw248. No abstract available. PMID 28338877
- [Background] Williamson T, Green ME, Birtwhistle R, Khan S, Garies S, Wong ST, Natarajan N, Manca D, Drummond N. Validating the 8 CPCSSN case definitions for chronic disease surveillance in a primary care database of electronic health records. Ann Fam Med. 2014 Jul;12(4):367-72. doi: 10.1370/afm.1644. PMID 25024246
- [Background] Queenan JA, Williamson T, Khan S, Drummond N, Garies S, Morkem R, Birtwhistle R. Representativeness of patients and providers in the Canadian Primary Care Sentinel Surveillance Network: a cross-sectional study. CMAJ Open. 2016 Jan 25;4(1):E28-32. doi: 10.9778/cmajo.20140128. eCollection 2016 Jan-Mar. PMID 27331051
- [Background] Coons MJ, Greiver M, Aliarzadeh B, Meaney C, Moineddin R, Williamson T, Queenan J, Yu CH, White DG, Kiran T, Kane JJ. Is glycemia control in Canadians with diabetes individualized? A cross-sectional observational study. BMJ Open Diabetes Res Care. 2017 Jun 8;5(1):e000316. doi: 10.1136/bmjdrc-2016-000316. eCollection 2017. PMID 28761645
- [Background] Morkem R, Williamson T, Patten S, Queenan JA, Wong ST, Manca D, Barber D. Trends in antidepressant prescribing to children and adolescents in Canadian primary care: A time-series analysis. Pharmacoepidemiol Drug Saf. 2017 Sep;26(9):1093-1099. doi: 10.1002/pds.4240. Epub 2017 Jun 8. PMID 28594077
- [Background] Greiver M, Williamson T, Barber D, Birtwhistle R, Aliarzadeh B, Khan S, Morkem R, Halas G, Harris S, Katz A. Prevalence and epidemiology of diabetes in Canadian primary care practices: a report from the Canadian Primary Care Sentinel Surveillance Network. Can J Diabetes. 2014 Jun;38(3):179-85. doi: 10.1016/j.jcjd.2014.02.030. Epub 2014 May 14. PMID 24835515
- [Background] Patton M. Qualitative evaluation and research methods. 2nd ed. Newbery Park, CA: Sage Publication; 1990.
- [Background] Sopcak N, Aguilar C, O'Brien MA, Nykiforuk C, Aubrey-Bassler K, Cullen R, Grunfeld E, Manca DP. Implementation of the BETTER 2 program: a qualitative study exploring barriers and facilitators of a novel way to improve chronic disease prevention and screening in primary care. Implement Sci. 2016 Dec 1;11(1):158. doi: 10.1186/s13012-016-0525-0. PMID 27906041
- [Background] Glaser B, Strauss A. The discovery of grounded theory: Strategies for qualitative research. New York: Aldine de Gruyter; 1967.
- [Background] Strauss A, Corbin J. Basics of qualitative research: Grounded theory procedures and techniques. Newbury Park, CA: Sage; 1990.
- [Background] Graham ID, Logan J, Harrison MB, Straus SE, Tetroe J, Caswell W, Robinson N. Lost in knowledge translation: time for a map? J Contin Educ Health Prof. 2006 Winter;26(1):13-24. doi: 10.1002/chp.47. PMID 16557505
- [Background] UTOPIAN Idea to Proposal Course (I2P). 2016; http://www.dfcm.utoronto.ca/utopian-idea-proposal-course-i2p.
- [Background] Grant A, Dreischulte T, Guthrie B. Process evaluation of the Data-driven Quality Improvement in Primary Care (DQIP) trial: case study evaluation of adoption and maintenance of a complex intervention to reduce high-risk primary care prescribing. BMJ Open. 2017 Mar 10;7(3):e015281. doi: 10.1136/bmjopen-2016-015281. PMID 28283493
- [Background] Helfrich CD, Li YF, Sharp ND, Sales AE. Organizational readiness to change assessment (ORCA): development of an instrument based on the Promoting Action on Research in Health Services (PARIHS) framework. Implement Sci. 2009 Jul 14;4:38. doi: 10.1186/1748-5908-4-38. PMID 19594942
- [Derived] Greiver M, Dahrouge S, O'Brien P, Manca D, Lussier MT, Wang J, Burge F, Grandy M, Singer A, Twohig M, Moineddin R, Kalia S, Aliarzadeh B, Ivers N, Garies S, Turner JP, Farrell B. Improving care for elderly patients living with polypharmacy: protocol for a pragmatic cluster randomized trial in community-based primary care practices in Canada. Implement Sci. 2019 Jun 6;14(1):55. doi: 10.1186/s13012-019-0904-4. PMID 31171011

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/49/NCT03689049/Prot_SAP_ICF_000.pdf